CLINICAL TRIAL: NCT03117166
Title: Effect of Intravenous Lidocaine, Used to Attenuate Pain With Propofol Injection, on Defibrillation Threshold Testing
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: multidisciplinary participation could not be overcome.
Sponsor: Drexel University College of Medicine (Other)
Responsible Party: Sponsor
Organization: Drexel University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 17283
Record Dates: First submitted 2011-05-24; First posted 2017-04-17 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Pain
Keywords: lidocaine implantation ICD
MeSH Terms: conditions — Pain | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lidocaine (Experimental): treatment arm
  Interventions: Drug: lidocaine
- Saline (Placebo Comparator): placebo arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: lidocaine — A one time bolus of lidocaine 0.5 mg/kg iv will be administered just prior to IV propofol injection,then successful defibrillation will be ascertained
  Arms: Lidocaine
Drug: Placebo — A control group will get an IV bolus of 0.9% NS just prior to IV bolus of propofol, then successful defibrillation will be ascertained
  Other Names: Saline
  Arms: Saline

SUMMARY:
The use of lidocaine, as an anesthetic drug, during implantation of an implantable cardioverter-defibrillator(ICD)will not result in a clinically significant alteration of the defibrillation threshold during ICD placement.

DETAILED DESCRIPTION:
Summary: The purpose is to observe the incidence of successful defibrillation on the first attempt during implantation of an implantable cardioverter-defibrillator (ICD) among patients who receive a standard dose of intravenous lidocaine (for attenuation of pain associated with propofol injection) versus patients who do not receive an intravenous lidocaine dose.

During implantation of an ICD, defibrillation threshold (DFT) testing is performed. DFT is calibrated as the lowest energy delivered by the ICD that will successfully terminate malignant arrhythmia. Lidocaine, a routine anesthetic agent, is also identified as an antiarrhythmic drug. Experimentally, lidocaine has been shown to increase thresholds during DFT' testing due to the drugs dual effect. The rationale behind this project is that the lidocaine may yield falsely elevated DFT, resulting in higher calibration of the ICD device. This alteration can affect ICD battery and overall ICD life. Comparisons between study groups may elucidate effects of IV lidocaine on DFT.

ELIGIBILITY:
Inclusion Criteria:

* Any person referred to the Hahnemann University Hospital Electrophysiology Laboratory for a clinically indicated ICD implant

Exclusion Criteria:

* Any person under the age of 18 years
* Inability to give an informed consent
* Allergy to lidocaine
* Receiving lidocaine treatment for pain or arrhythmia
* Contraindication for DFT testing
* Not consenting for DFT testing
* Receiving energy other than 10-12.5 joules as initial DFT test
* Implant of ICD on the right side
* DFT not planned to be performed during ICD implant
* Epicardial placement of ICD leads
* Use of single coil ICD lead
* Subpectoral ICD implantation
* Cephalic cutdown used for central venous access
* Require more than 3mg/kg of 1% SQ lidocaine for local anesthesia
* Pregnant women or prisoners

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Incidence of successful defibrillation on first attempt with 10-12 joules. | Through study completion but no longer than 1 year
  These patients will receive a standard dose of intravenous lidocaine (for attenuation of pain associated with propofol injection) versus patients who do not receive an intravenous lidocaine dose. Outcome is to have a success defibrillation within the first attempt.

SECONDARY OUTCOMES:
Incidence of failure to defibrillate at higher energy levels. | Through study completion but no longer than 1 year
  This outcome occurs when research team fails to defibrillate on any attempt.
Defibrillation threshold (DFT) for subjects who fail to defibrillate at the initial 10-12 joules. | Through study completion but no longer than 1 year
  This outcome occurs when research team fails to defibrillate on first attempt.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Chambers, Principal Investigator — Drexel
Locations (1):
- Hahnemann University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No